CLINICAL TRIAL: NCT05990140
Title: The Effect of Peppermint Flavored Mouthwash Applied to Patients in the First 30 Days After Bariatric Surgery on Nausea-Vomiting, Anxiety and Biochemical Parameters
Brief Title: The Effect of Peppermint Flavored Mouthwash Applied to Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Vesile Eskici Ilgin, Principal Investigator, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Vesile23
Record Dates: First submitted 2023-07-19; First posted 2023-08-14 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Postoperative Complications
Keywords: nausea-vomiting; anxiety; nurse; Biochemical Parameters
MeSH Terms: conditions — Postoperative Complications; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Consent of all patients will be obtained the night before surgery. Biochemical parameter levels and state trait anxiety scale and apfel risk scale will be recorded.
  As it will be difficult for the experimental group to be oriented while giving mouthwash training after the surgery, mouthwash training will be given at a time when it is available the night before the operation. State anxiety scale, visual comparison scale and nausea and vomiting effect scale will be administered before discharge (approximately 48 hours). After discharge, he will continue to gargle in the same way 3 times a day. At the end of the first week, all patients will be called by the researcher and the state anxiety scale, visual comparison scale and nausea and vomiting effect scale shared on the digital environment will be filled and recorded. This process will continue for 4 weeks. In the last measurement, visual comparison scale, nausea vomiting and state trait anxiety scale will also be filled.
  Interventions: Other: peppermint flavored mouthwash
- Control (No Intervention): Consent of all patients will be obtained the night before surgery. Biochemical parameter levels and state trait anxiety scale and apfel risk scale will be recorded.
  The state anxiety scale, visual comparison scale and nausea and vomiting effect scale will be administered to the control group before they are discharged (approximately at the 48th hour). At the end of the first week, all patients will be called by the researcher, and the state anxiety scale, visual comparison scale and nausea and vomiting effect scale will be filled and recorded. This process will continue for 4 weeks. In the last measurement, visual comparison scale, nausea vomiting and state trait anxiety scale will also be filled. At the end of the first month, the biochemical parameters taken during the routine hospital control will be recorded.

INTERVENTIONS:
Other: peppermint flavored mouthwash — The Effect of Peppermint Flavored Mouthwash Applied to Patients in the First 30 Days After Bariatric Surgery on Nausea-Vomiting, Anxiety and Biochemical Parameters
  Arms: Experimental

SUMMARY:
Treatment of obesity consists of diet/lifestyle modification and bariatric surgery consisting of several procedures. One of the most common complications in the early period after bariatric surgery is nausea and vomiting due to the reduction of gastric capacity. According to the guidelines of the American Society of Metabolic and Bariatric Surgery (ASMBS), acid-base disorders, electrolyte abnormalities (especially calcium, potassium, magnesium, sodium and phosphorus deficiency), insufficiency of fat-soluble vitamins (ADEK), folic acid, iron, thiamine after bariatric surgery. and B12 deficiency etc. On the other hand, anxiety after bariatric surgery is also an important problem.

It is possible to reduce nausea and vomiting by stimulating the vagal nerve. Gargling, laughing, singing loudly, etc. The movements stimulate the vagus nerve by activating the muscles behind the larynx, and the vagus nerve prevents nausea and vomiting by simulating the gastrointestinal tract. With the activation of the diaphragm; The vagus nerve is stimulated, the parasympathetic nervous system is activated and cortisol production decreases, reducing stress and anxiety. The peppermint plant, which is widely used in our country, is also used as a relief in cases such as nausea, stomachache, and colds. It is expected that the nurse, who is a member of the multidisciplinary team, will be able to properly define the surgical risks and comorbidities associated with the clinical status of obesity in patients who have undergone bariatric surgery and to apply the necessary interventions.

ELIGIBILITY:
Inclusion Criteria:

1. Be between the ages of 18-65
2. Having had bariatric surgery
3. Absence of communication barriers
4. Volunteering to participate in research
5. Mental well-being

Exclusion Criteria:

1. Presence of major depression or psychosis
2. Having a communication barrier
3. Being transferred to another unit
4. Leaving work voluntarily

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-08-15 (Estimated); Primary Completion 2024-05-12 (Estimated); Study Completion 2024-07-15 (Estimated)

PRIMARY OUTCOMES:
State-Trait Anxiety Inventory | up to 1 month
  This inventory consists of two separate sections. consists of 40 questions in total. General temperament of the person in 20 questions in the continuous section While the state is evaluated, how the person feels at that moment is evaluated in the state section. Continually Anxiety is an individual's tendency to experience anxiety. State anxiety is the stressful situation in which the individual is It is the subjective fear felt by the situation. While it rises when the stress is intense, the stress In cases where the level of anxiety decreases, the State-Trait Anxiety Inventory score decreases. Inventory While filling, one of the 4 options is preferred; scores are added together and high scores are shows anxiety levels
Nausea Vomiting Visual Comparison Scale | up to 1 month
  It is a scale that evaluates the severity of nausea of the participants on a 10-centimeter ruler with "0" on the left end, no nausea at all, and "100" on the right end as the most severe nausea (unbearable nausea).
Determination of Levels of Biochemical Parameters in Blood | up to 1 month
  Laboratory results obtained routinely in the hospital where the study will be conducted will be used.

CONTACTS AND LOCATIONS:
Overall Officials: Vesile Eskici İlgin, Dr, Principal Investigator — Ataturk University

IPD SHARING:
Plan to Share IPD: No